CLINICAL TRIAL: NCT04020978
Title: Pilot Study Using Parametric PET to Assess Early Treatment Response to Targeted Therapy for Genitourinary Cancer (GUC)
Brief Title: Parametric PET of Genitourinary Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1374902
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Genitourinary Cancer
Keywords: Functional Imaging; Dynamic PET; tracer kinetic modeling; treatment response
MeSH Terms: conditions — Urogenital Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with GUC (Other): Each patient with GUC will first undergo an X-ray CT scan for attenuation correction purpose. After that, 10 mCi 18F-Fludeoxyglucose (18F-FDG) will be injected into the patient through the IV in a period of 10 seconds. The PET scan commences 10 seconds before the FDG injection and lasts for 60 minutes. After the PET scan, the patient gets off the scanner. One blood sample (10cc) will be drawn using a butterfly method with the time recorded.
  Interventions: Diagnostic Test: Parametric PET/CT

INTERVENTIONS:
Diagnostic Test: Parametric PET/CT — Each patient will undergo a dynamic F18-FDG PET/CT scan at baseline and 2-week post therapy.

SUMMARY:
Metastatic kidney cancer is usually treated with targeted therapy or immunotherapy which is costly and has low response rate. The current standard care is to perform anatomical imaging studies after a few cycles (months) of treatment to evaluate response. This approach exposes many patients to highly toxic, high expensive treatment without any benefit for months and delays initiation of other effective therapies. The goal of this study is to evaluate a parametric PET method that potentially identify response and assess drug efficacy with a few days to weeks of treatment.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is one of the top ten cancer types in the US. One-third of RCCs are metastatic and associated with a poor 5-year survival rate of 8%. Metastatic RCC is usually treated with targeted therapy or immunotherapy which is costly (>$10,000 per month) and has low response rate (<30%). Effective identification of the most appropriate drugs for a patient relies on noninvasive imaging to assess early response to the drugs. However, current practice by anatomical imaging such as computed tomography (CT) or magnetic resonance imaging (MRI) can only assess the response at two months after initialing targeted therapy. This approach exposes many patients to highly toxic, high expensive treatment without any benefit for months and delays initiation of other effective therapies.

The investigators hypothesize that functional perfusion imaging by positron emission tomography (PET) can enable RCC response assessment as early as at 1-2 weeks given that RCC is highly related to angiogenesis and most targeted drugs for RCC are antiangiogenic. However, clinical options for functional renal imaging are very limited. While dynamic contrast-enhanced CT or MRI can be used for perfusion imaging, their use is restricted because 30% of RCC patients have chronic kidney diseases with renal dysfunction and are at higher risk for contrast-induced nephropathy and nephrogenic systemic fibrosis. Existing PET radiotracers (e.g., 15O-water) for perfusion imaging are short-lived and generally unavailable for clinical use. This project explores parametric PET perfusion imaging using the widely accessible 18F-fluorodeoxyglucose (FDG). 18F-FDG PET is conventionally used for metabolic imaging and has been rarely used for imaging kidneys because physiological excretion of 18F-FDG into renal pelvis contaminates image quality for renal tumor assessment. The investigators explore the potential of the metabolic radiotracer 18F-FDG for perfusion imaging by employing four-dimensional (4D: 3D space plus 1D time) dynamic scanning and tracer kinetic modeling, leading to parametric imaging of FDG perfusion kinetics without being affected by 18F-FDG excretion. The parametric PET method can potentially identify RCC response and assess drug efficacy with 1-2 weeks of treatment as compared to 2 months by current anatomical imaging methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed GUC. For those patients whose primary kidney cancer is removed, they must have index metastatic cancer lesion(s) within the PET field of view for 18F-FDG parametric PET/CT analysis to determine response.
* Patients are scheduled for targeted cancer therapy, including sunitinib, pazopanib, cabozantinib, everolimus, and others.
* Ability to understand and willingness to sign an informed consent form.
* Ability to adhere to the study visit schedule and other protocol requirements.
* Men and women ≥21 years of age.
* Life expectancy ≥ 6months.
* Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for ≥1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Or, female subjects of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the first drug administration.
* Male and female subjects who agree to use highly effective method of birth control (e.g., implants, injectables, birth control pills with two hormones, intrauterine devices [IUDs], complete abstinence or sterilized partner, and female sterilization) and a barrier method (e.g., condoms, vaginal ring, sponge, etc.) during the period of therapy and for 90 days after the last dose of drug.
* For the minority cohort, subject must be a member of a Federally recognized racial/ethnic minority population to include: African Americans or Black; Native American; Alaska Native; Native Hawaiian or other Pacific Islander; Asian American; Hispanic or Latino. This will be verified through self-reporting by the subject.

Exclusion Criteria:

* Pregnant or lactating women.
* Any condition that would prohibit the understanding or rendering of informed consent.
* Any medical condition including additional malignancies, laboratory abnormalities, or psychiatric illness that would prevent the subject from participating and adhering to study related procedures.
* Prior treatment with any investigational drug within the previous 4 weeks
* Unable to lie supine for 1-hour imaging with PET
* Prisoners

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in blood flow | Two weeks
  Tumor blood flow in the unit of mL/min/g will be derived from early-dynamic FDG-PET with tracer kinetic modeling. The change between baseline and follow-up scans will be calculated.
Changes in blood volume | Two weeks
  Tumor blood volume fraction in percentage will be derived from early-dynamic FDG-PET with tracer kinetic modeling. The change between baseline and follow-up scans will be calculated.

SECONDARY OUTCOMES:
Correlation with tumor anatomical response | Two months
  Correlation between the functional changes measured by parametric PET/CT at two weeks with anatomical size change measured by standard CT or MRI at two months.

OTHER OUTCOMES:
Inclusion of Minority Cohort | One year after treatment
  Inclusion of subjects of various race and/or ethnicity to ensure findings can be generalizable to the entire population and to gather information about differences by race and/or ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Guobao Wang, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No